CLINICAL TRIAL: NCT02428634
Title: The Program SI! for Cardiovascular Health Promotion for Elementary Students Aged 6 to 11: a Cluster Randomized Trial
Brief Title: The Program SI! for Cardiovascular Health Promotion at Elementary School
Acronym: PSIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Science, Health and Education, Spain (Other)
Collaborators: Fondation Daniel & Nina Carasso (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHE-002-SI
Record Dates: First submitted 2015-04-08; First posted 2015-04-29 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular health promotion; Children; School intervention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Program SI! for Elementary 6 levels (Experimental): The core intervention comprises classroom activities grouped in healthy challenges (about diet, physical activity, human body and heart, and emotions management) distributed across the different levels and implemented by the corresponding teachers. All the materials, formal training and a teaching guide are provided to the school staff by the SHE Foundation. Families receive family-challenges and key messages about their children's health. The school environment is intervened mainly through an annual Healthy Fair. The intervention is implemented during all the elementary levels (PSIE13+PSIE46).
  Interventions: Behavioral: PSIE13; Behavioral: PSIE46
- Normal curriculum (No Intervention): The schools on the control group keep their normal curriculum and don't join any school program about health until the end of the study.
- Program SI! for Elementary first levels (Experimental): The core intervention comprises classroom activities grouped in healthy challenges (about diet, physical activity, human body and heart, and emotions management) distributed across the different levels and implemented by the corresponding teachers. All the materials, formal training and a teaching guide are provided to the school staff by the SHE Foundation. Families receive family-challenges and key messages about their children's health. The school environment is intervened mainly through an annual Healthy Fair. To evaluate the effects of different exposures to the program, the intervention is implemented in the first three levels (PSIE13).
  Interventions: Behavioral: PSIE13
- Program SI! for Elementary last levels (Experimental): The core intervention comprises classroom activities grouped in healthy challenges (about diet, physical activity, human body and heart, and emotions management) distributed across the different levels and implemented by the corresponding teachers. All the materials, formal training and a teaching guide are provided to the school staff by the SHE Foundation. Families receive family-challenges and key messages about their children's health. The school environment is intervened mainly through an annual Healthy Fair. To evaluate the effects of different exposures to the program, the intervention is implemented in the last three levels (PSIE46).
  Interventions: Behavioral: PSIE46

INTERVENTIONS:
Behavioral: PSIE13 — The Program SI! is implemented from 1st to 3rd grade of Elementary. A total of 40 hours of intervention on 1st and 2nd grade and 30 hours on 3rd grade has been established as the minimum intervention per year.
  Arms: Program SI! for Elementary 6 levels; Program SI! for Elementary first levels
Behavioral: PSIE46 — The Program SI! is implemented from 4th to 6th grade of Elementary. A total of 30 hours of intervention has been established as the minimum intervention per year.
  Arms: Program SI! for Elementary 6 levels; Program SI! for Elementary last levels

SUMMARY:
The objective of the study is to evaluate the effects of Program SI! for Elementary in different times of exposure for childrens and their immediate environment (teachers and parents). For this purpose, 48 public schools from the Community of Madrid-South Area (Spain) were randomly assigned to Program SI! during 3 or 6 academic years (intervention group) or keep their normal curriculum (control group). The main outcome is 3-year, and 6-year changes from baseline of questionnaire scoring of children, their parents and teachers in regards to a healthy lifestyle. For children were included 3-year, and 6-year changes of cardiovascular markers derived from blood pressure and anthropometry.

DETAILED DESCRIPTION:
The Program SI! is a multilevel school-based intervention integrating four cardiovascular health-related components (diet, physical activity, human body and emotions management). Since the Program SI! for preschoolers has shown good results in improving healthy lifestyle habits in children aged 3 to 5 years, the investigators have developed the Program SI! for Elementary addressed to children from 6 to 11 years. The objective of the study is to evaluate the effects of Program SI! for Elementary in different times of exposure for childrens and their immediate environment (teachers, parents and school). In the Community of Madrid-South Area (Spain), 48 public schools from were randomly assigned to Program SI! for Elementary during 3 or 6 academic years (intervention group) or keep their normal curriculum (control group). The main outcome is 3-year, and 6-year changes from baseline of questionnaire scoring of children, and the secondary outcome is 3-year, and 6-year changes from baseline of questionnaire scoring of their parents and teachers in regards to a healthy lifestyle, as well as changes in the school environment. For children were included 3-year, and 6-year changes of cardiovascular markers derived from blood pressure and anthropometry (weight, height, waist circumference and skinfold thickness). The Program SI! for Elementary is designed for different exposures in a sample of schools never intervened to asses when the intervention has the most effectiveness. Besides, as some schools involved in the preschool study continues the Program SI! for Elementary, the investigators can be able to evaluate the impact of the Program SI! in different school stages, concluding how children keep the adoption of healthy behaviors from early in life.

ELIGIBILITY:
Inclusion Criteria:

* Children from public schools with canteen services located in the South Madrid Area of Education, having from 1st to 6th grades and at least two classrooms in 1st grade.

Exclusion Criteria:

* The coordination team of the SHE Foundation establishes the adherence criteria and the schools not reaching the minimum considered can be excluded. Questionnaires scoring from students with special educational needs will be excluded from the analysis of questionnaires, as well as repeat students.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1770 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Difference between control and intervention groups in the mean change in questionnaire's scoring from baseline to 3-year and 6-year intervention for children. | 3-year, and 6-year changes from baseline of questionnaire scoring for children
  To evaluate children's lifestyle we use a specific questionnaire about knowledge, attitudes and habits in relation to the four components of Program SI! for Elementary (diet, physical activity, body and heart, and emotions management) (article under revision). A trained team of psychologist applies the children's questionnaires at the school.
Cardiovascular health markers (blood pressure, height, weight, waist circumference and triceps and subscapular skinfold thickness) of children from baseline to 3-year and 6-year intervention. | 3-year, and 6-year changes from baseline on cardiovascular health markers of children
  To evaluate the impact of the Program SI! for Elementary in cardiovascular health markers of children blood pressure and some anthropometric parameters are measured (height, weight, waist circumference and triceps and subscapular skinfold thickness) under standardized protocol developed in previous studies (Santos-Beneit et al. 2014).

SECONDARY OUTCOMES:
Difference between control and intervention groups in the mean change in questionnaire's scoring from baseline to post-intervention for families. | 3-year, and 6-year changes from baseline of questionnaire scoring for families
  The family's habits are evaluated through a specific questionnaire related to key messages for families provided by the Program SI! for Elementary and some general questions about tobacco use and health status (article under revision) and stress perception (Remor 2006). Also in the questionnaire for families are included some questions about their son or daughter's habits (Serra-Majem et al 2004, Goodman 1997, Encuesta Nacional de Salud 2011/2012).
Difference between control and intervention groups in the mean change in questionnaire's scoring from baseline to post-intervention for teachers | 3-year, and 6-year changes from baseline of questionnaire scoring for teachers
  The lifestyle of the teachers is evaluated measuring adherence to the Mediterranean lifestyle (Sotos-Prieto et al. 2014) and questions about stress perception (Remor 2006).
Difference between control and intervention groups in the mean change in questionnaire's scoring from baseline to post-intervention for school environment | 3-year, and 6-year changes from baseline of questionnaire scoring for school environment
  The school environment is evaluated through questions related to the recommendations provided in the Program SI! for Elementary intervention as avoid eating commercially prepared baked foods at school.

CONTACTS AND LOCATIONS:
Overall Officials: Valentín Fuster, MD, PhD, Study Chair — Chairman of the Foundation for Science, Health and Education
Locations (1):
- Foundation for Science, Health and Education, Madrid, Spain

REFERENCES:
- [Background] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Sotos-Prieto M, Moreno-Franco B, Ordovas JM, Leon M, Casasnovas JA, Penalvo JL. Design and development of an instrument to measure overall lifestyle habits for epidemiological research: the Mediterranean Lifestyle (MEDLIFE) index. Public Health Nutr. 2015 Apr;18(6):959-67. doi: 10.1017/S1368980014001360. Epub 2014 Jul 15. PMID 25025396
- [Background] Remor E. Psychometric properties of a European Spanish version of the Perceived Stress Scale (PSS). Span J Psychol. 2006 May;9(1):86-93. doi: 10.1017/s1138741600006004. PMID 16673626
- [Background] Santos-Beneit G, Sotos-Prieto M, Pocock S, Redondo J, Fuster V, Penalvo JL. Association between anthropometry and high blood pressure in a representative sample of preschoolers in madrid. Rev Esp Cardiol (Engl Ed). 2015 Jun;68(6):477-84. doi: 10.1016/j.rec.2014.09.002. Epub 2014 Dec 6. PMID 25487220
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Santos-Beneit G, Bodega P, de Miguel M, Rodriguez C, Carral V, Orrit X, Haro D, Carvajal I, de Cos-Gandoy A, Penalvo JL, Gomez-Pardo E, Oliva B, Ibanez B, Fernandez-Alvira JM, Fernandez-Jimenez R, Fuster V. Rationale and design of the SI! Program for health promotion in elementary students aged 6 to 11 years: A cluster randomized trial. Am Heart J. 2019 Apr;210:9-17. doi: 10.1016/j.ahj.2018.12.011. Epub 2019 Jan 8. PMID 30716509
- See also: Encuesta Nacional de Salud España 2011/2012 — https://www.mscbs.gob.es/estadEstudios/estadisticas/encuestaNacional/encuesta2011.htm
- See also: Program SI! website — http://programasi.org/es/